CLINICAL TRIAL: NCT03820947
Title: Global, Post-Market, Prospective, Multi-Center, Randomized Controlled Trial of the VenaSeal™ Closure System vs. Surgical Stripping or Endothermal Ablation (ETA) for the Treatment of Early & Advanced Stage Superficial Venous Disease
Brief Title: VenaSeal Spectrum: Global Post-Market Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Follow-up of the VenaSeal vs. Endothermal Ablation and Venous Leg Ulcer studies was concluded early due to increased evidence of safety and effectiveness of VenaSeal in published literature and to reduce burden to investigators and sites.
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDT18034
Record Dates: First submitted 2019-01-08; First posted 2019-01-29 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Venous Reflux
Keywords: Venous reflux; Venous leg ulcer; Varicose Veins; Chronic Venous Insufficiency; VenaSeal; Endothermal Ablation; Surgical Stripping; Radiofrequency Ablation; Laser Ablation; Great Saphenous Vein; Small Saphenous Vein; Anterior Accessory Saphenous Vein
MeSH Terms: conditions — Varicose Ulcer; Varicose Veins | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Randomized study VenaSeal™ System versus Endothermal Ablation (ETA): VenaSeal™ System (Experimental): CEAP 2-5 subjects will be randomized to VenaSeal™ System vs. ETA
  Interventions: Device: VenaSeal™ System
- Randomized study VenaSeal™ System versus Endothermal Ablation (ETA): ETA (Active Comparator): CEAP 2-5 subjects will be randomized to VenaSeal™ System vs. ETA
  Interventions: Device: Endothermal Ablation (ETA)
- Randomized study VenaSeal™ System versus Surgical Stripping: VenaSeal™ System (Experimental): CEAP 2-5 subjects will be randomized to VenaSeal™ System vs. Surgical Stripping
  Interventions: Device: VenaSeal™ System
- Randomized study VenaSeal™ System versus Surgical Stripping: Surgical Stripping (Active Comparator): CEAP 2-5 subjects will be randomized to VenaSeal™ System vs. Surgical Stripping
  Interventions: Procedure: Surgical Stripping
- Single arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System (Experimental): CEAP 6 active leg ulcer subjects will not be randomized to a comparator, all subjects will be treated with VenaSeal™ System
  Interventions: Device: VenaSeal™ System

INTERVENTIONS:
Device: VenaSeal™ System — The VenaSeal™ System is the non-tumescent, non-thermal, non-sclerosant device that uses a proprietary medical adhesive delivered endovenously to close the vein.
  Arms: Randomized study VenaSeal™ System versus Endothermal Ablation (ETA): VenaSeal™ System; Randomized study VenaSeal™ System versus Surgical Stripping: VenaSeal™ System; Single arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Device: Endothermal Ablation (ETA) — ETA includes EVLA that uses laser or RFA that uses radiofrequency heating to close the vein. Heat is applied in both EVLA and RFA therapies to close the vein.
  Subject can be treated with either EVLA or RFA if randomized to ETA arm per site's standard practice.
  Other Names: Endovenous laser ablation (EVLA); Radiofrequency ablation (RFA)
  Arms: Randomized study VenaSeal™ System versus Endothermal Ablation (ETA): ETA
Procedure: Surgical Stripping — Surgical stripping involves stripping (removal) of the diseased vein via surgical procedures.
  Arms: Randomized study VenaSeal™ System versus Surgical Stripping: Surgical Stripping

SUMMARY:
Global, Post-Market, Prospective, Multi-Center, Randomized Controlled Trial of the VenaSeal™ Closure System vs. Surgical Stripping or Endothermal Ablation (ETA) for the Treatment of Early and Advanced Stage Superficial Venous Disease

DETAILED DESCRIPTION:
The study is designed with two randomized studies and one single arm study.

Two randomized studies are for CEAP 2-5 subjects:

1. VenaSeal vs. Surgical Stripping Study (outside of the United States only)
2. VenaSeal vs. ETA Study

The single arm study is for CEAP 6 subjects with active venous leg ulcers (VLU):

1. VLU Study

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age
2. Patient has venous reflux in superficial truncal vein(s) (e.g., GSV, SSV, accessory saphenous veins) with CEAP 2 (symptomatic) or CEAP 3, 4a, 4b, 5, 6, appropriate for treatment, as confirmed by Duplex Ultrasound (DUS)
3. Eligibility for treatment:

   * VenaSeal vs ETA Study: Patient is eligible for treatment with the VenaSeal™ system and ETA
   * VenaSeal vs Surgical Stripping Study: Patient is eligible for treatment with the VenaSeal™ system and surgical stripping
   * VLU Study: patients should be eligible for treatment with the VenaSeal™ system
4. Treatable refluxing segment of target vein(s) 10 cm in length or longer
5. Patient has a target vein diameter of ≥3 mm throughout the intended treated segment of the target vein as measured by DUS while patient is standing
6. Patient is willing and capable of complying with specified follow-up evaluations at the specified times
7. Patient has an ability to understand the requirements of the study and to provide informed consent

Exclusion Criteria:

1. Patient has a known history of allergic sensitivities (including but not limited to cyanoacrylate adhesives), or any other condition, which in the opinion of the investigator may make the patient more susceptible to cyanoacrylate adhesive hypersensitivity
2. Patient has known deep vein obstruction in the target limb, as identified by the site's standard of care
3. Patient has abnormal pulse exam or ABI <0.8
4. Patient has acute superficial thrombophlebitis
5. Patient requires any non-target vein treatments in the contralateral or ipsilateral limb, or any other surgical procedure up tp 30 days pre-procedure and through 3 months post-procedure
6. Patient has any co-morbid conditions, which in the investigator's opinion may interfere with the patient's compliance with study visits and procedures, or may confound interpretation of study data (e.g., congestive heart failure Class III and IV, non-ambulatory patients, severe hepatic dysfunction, life expectancy < 1 year)
7. IFU contraindications:

   * VenaSeal vs. ETA Study: Patient has VenaSeal™ system and/or ETA product's IFU contraindication(s)
   * VenaSeal vs Surgical Stripping Study: Patient has surgical stripping and/or VenaSeal™ system IFU contraindication(s)
   * VLU Study: Patient has VenaSeal™ system IFU contraindication(s)
8. Patient is non-ambulatory
9. Patient is a female of childbearing potential who may be pregnant or breastfeeding at the time of the index procedure
10. Patient belongs to a vulnerable population per investigator's judgment or patient has any kind of disorder that compromises his/her ability to give written informed consent and/or to comply with study procedures
11. Patient is currently participating in an investigational drug or device study when the data collected could be conflicting or biased due to participation in another study
12. Patient has documented COVID-19 infection currently or within the past 3 months. Patient is not completely recovered from past COVID-19 infection, per physician's discretion.
13. VLU Study: Patient has target ulceration identified to be of non-venous etiology, as confirmed by the independent core laboratory
14. VLU Study: Patient has target circumferential ulceration that cannot be captured in a single photograph (any ulcer curvature around the leg that goes out of sight)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2025-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Gibson, MD, Principal Investigator — Lake Washington Vascular, US; Manjit Gohel, MD, Principal Investigator — Addenbrooke's Hospital, UK
Locations (32):
- United States (12):
  - Yavapai Regional Medical Center, Prescott Valley, Arizona
  - PIMA Heart and Vascular, Tucson, Arizona
  - Valley Vascular Surgical Associates, Fresno, California
  - Vascular Care Connecticut, Darien, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Vascular Care Group, Wellesley, Massachusetts
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Orion Medical, Houston, Texas
  - Lake Washington Vascular, Bellevue, Washington
- Australia (2):
  - Sunshine Coast University Hospital, Birtinya
  - Wollongong Hospital, Wollongong
- East Toronto Vascular Clinic, Toronto, Ontario, Canada
- France (3):
  - CHU Dijon Bourgogne, Dijon, DIjon Cedex
  - Clinique du Parc, Lyon
  - Clinique Pasteur, Toulouse
- Praxis fur Innere Medizin und Gefäβkrankheiten, Halle, Germany
- Italy (2):
  - Ospedale Fatebenefratelli e Oftalmico, Milan
  - Azienda Ospedaliera di Padova Ospendale Sant' Antonio, Padua
- Rijnstate - Locatie Arnhem, Arnhem, Netherlands
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
- Spain (2):
  - Complejo Hospitalario Universitario Granada (Hospital Campus de la Salud), Granada
  - Sanitas Hospital Universitario La Zarzuela, Madrid
- United Kingdom (4):
  - Bedfordshire Hospitals NHS Foundation Trust, Bedford
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital, Cambridge
  - West London Vascular and Interventional Centre, Harrow
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA: CEAP 2-5 subjects will be randomized to VenaSeal™ System vs. ETA
  Endothermal Ablation (ETA): ETA includes EVLA that uses laser or RFA that uses radiofrequency heating to close the vein. Heat is applied in both EVLA and RFA therapies to close the vein.
  Subject can be treated with either EVLA or RFA if randomized to ETA arm per site's standard practice.
Period: Overall Study
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Started | 136 | 139 | 53 | 53 | 125
Completed (12 month is primary endpoint timepoint) | 115 | 104 | 43 | 39 | 87
Not Completed | 21 | 35 | 10 | 14 | 38
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 6 | 10 | 3 | 8 | 5
Not completed — Procedure Not Attempted | 0 | 2 | 1 | 0 | 0
Not completed — Other Exit | 1 | 3 | 3 | 3 | 0
Not completed — Follow-up Not Done | 10 | 13 | 2 | 3 | 12
Not completed — Death | 0 | 0 | 0 | 0 | 9
Not completed — Lost to Follow-up | 4 | 6 | 0 | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System | Total
Number analyzed (Participants) | 136 | 139 | 53 | 53 | 125 | 506
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Overall Number of Baseline Participants is the number of ITT. The number analyzed participants is the number with available data for this baseline measure.
  years
    number analyzed (Participants) | 131 | 130 | 50 | 49 | 125 | 485
    (all) | 57.0 (13.20) | 57.2 (13.70) | 60.3 (14.39) | 61.5 (12.96) | 67.9 (14.76) | 60.7 (14.52)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Overall Number of Baseline Participants is the number of ITT. The number analyzed participants is the number with available data for this baseline measure.
  Participants
    Female: number analyzed (Participants) | 131 | 130 | 50 | 49 | 125 | 485
    Female | 91 | 78 | 29 | 33 | 48 | 279
    Male: number analyzed (Participants) | 131 | 130 | 50 | 49 | 125 | 485
    Male | 40 | 52 | 21 | 16 | 77 | 206
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Overall Number of Baseline Participants is the number of ITT. The number analyzed participants is the number with available data for this baseline measure.
  Race is not allowed to be collected per local laws or regulations in the following countries: France, Germany, Italy, The Netherlands, Spain, United Kingdom. Subjects could report more than one races; therefore the column total might be more than the study arm total.
  Participants
    Not reportable per local laws or regulations: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Not reportable per local laws or regulations | 67 | 69 | 7 | 4 | 55 | 202
    Subject declines to answer: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Subject declines to answer | 0 | 3 | 0 | 0 | 0 | 3
    Unknown: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Unknown | 0 | 0 | 0 | 0 | 3 | 3
    Black or African American: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Black or African American | 1 | 1 | 0 | 0 | 3 | 5
    Chinese: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Chinese | 0 | 0 | 0 | 0 | 0 | 0
    Japanese: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Japanese | 0 | 0 | 0 | 0 | 0 | 0
    Korean: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Korean | 13 | 14 | 38 | 41 | 0 | 106
    Native American or Alaska Native: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Native American or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific islander: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Native Hawaiian or Other Pacific islander | 0 | 1 | 0 | 0 | 0 | 1
    White: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    White | 50 | 42 | 5 | 3 | 63 | 163
    Other Asian: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Other Asian | 0 | 1 | 0 | 0 | 1 | 2
    Other: number analyzed (Participants) | 131 | 130 | 50 | 48 | 125 | 484
    Other | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Population: Overall Number of Baseline Participants is the number of ITT. The number analyzed participants is the number with available data for this baseline measure.
  kg/m2
    number analyzed (Participants) | 131 | 130 | 50 | 47 | 125 | 483
    (all) | 26.4 (4.93) | 27.9 (5.77) | 25.8 (5.77) | 24.2 (3.41) | 32.4 (9.35) | 28.1 (7.08)
CEAP: Clinical, Etiological, Anatomical, and Pathophysiological Classification [Count of Participants; unit: Participants] — Clinical Classification per 2004 guidelines C0: no visible or palpable signs of venous disease C1: telengiectasies or reticular veins C2: variose veins C3: edema C4a: pigmentation and eczema C4b: lipodermatosclerosis and atrophie blanche C5: healed venous ulcer C6: active venous ulcer Higher score means more advanced venous disease progression
  Participants
    C0 | 0 | 0 | 0 | 0 | 0 | 0
    C1 | 0 | 0 | 0 | 0 | 0 | 0
    C2 | 43 | 48 | 22 | 23 | 0 | 136
    C3 | 61 | 53 | 17 | 18 | 0 | 149
    C4a | 28 | 25 | 12 | 9 | 0 | 74
    C4b | 4 | 4 | 1 | 2 | 0 | 11
    C5 | 0 | 9 | 1 | 1 | 0 | 11
    C6 | 0 | 0 | 0 | 0 | 125 | 125

OUTCOME MEASURES:

1. Primary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Primary Endpoint: Peri-procedural Patient Satisfaction as Measured by a Validated, Patient-centered Venous Treatment Satisfaction Questionnaire (VenousTSQe) at 30 Days.
Description: Measured by a validated, patient-centered venous treatment satisfaction questionnaire - early (VenousTSQe).
  Total score ranges from 0-36, and a higher score means a higher peri-procedural venous treatment satisfaction.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 123 | 119
score on a scale | 30.8 (4.22) | 29.6 (4.73)

2. Primary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Primary Endpoint: Peri-procedural Patient Satisfaction as Measured by a Validated, Patient-centered Venous Treatment Satisfaction Questionnaire (VenousTSQe) at 30 Days.
Description: as for outcome 1
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 46 | 43
score on a scale | 29.3 (4.94) | 25.0 (6.24)

3. Primary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Primary Endpoint: Patient Satisfaction as Measured by a Validated, Patient-centered Venous Treatment Satisfaction Questionnaire (VenousTSQs) at 30 Days.
Description: Measured by a validated, patient-centered venous treatment satisfaction questionnaire - status (VenousTSQs).
  Total score ranges from 0-36, and a higher score means a higher venous treatment satisfaction.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 125 | 115
score on a scale | 31.8 (5.12) | 32.1 (4.95)

4. Primary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Primary Endpoint: Patient Satisfaction as Measured by a Validated, Patient-centered Venous Treatment Satisfaction Questionnaire (VenousTSQs) at 30 Days.
Description: as for outcome 3
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 46 | 43
score on a scale | 30.1 (6.39) | 28.3 (5.58)

5. Primary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Primary Endpoint: Elimination of Clinically Relevant Superficial Truncal Disease in Each Target Vein at the Time of Index Procedure.
Description: Elimination of clinically relevant superficial truncal disease in each target vein at the time of index procedure as measured by the percentage of target vein length successfully treated.
Time Frame: Post Index procedure, on the day of the procedure immediately following treatment
Population: Target Veins based measurement. Number of units analyzed corresponds to the number of target veins with available data.
Measure: Mean (Standard Deviation); unit: % of vein length
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 130 | 126
Number analyzed (Target Veins) | 137 | 130
% of vein length | 92.4 (13.40) | 91.1 (11.85)

6. Primary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Primary Endpoint: Elimination of Clinically Relevant Superficial Truncal Disease in Each Target Vein at the Time of Index Procedure.
Description: as for outcome 5
Time Frame: Post Index procedure, on the day of the procedure immediately following treatment
Population: Target Veins based measurement. Number of units analyzed units corresponds to number of target veins with available data.
Measure: Mean (Standard Deviation); unit: % of vein length
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
Number analyzed (Target Veins) | 49 | 44
% of vein length | 69.9 (19.93) | 68.2 (25.82)

7. Primary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Primary Endpoint: Time to Ulcer Healing, Calculated Through Healing Confirmation and Verified by an Independent Core Laboratory Through 12 Months.
Description: Time to ulcer healing reported by using the cumulative incidence probability estimate of the event happening at 12 months, expressed as a percentage. The data values below represent the cumulative incidence probability as a percentage of participants with ulcer healing through 12 months.
Time Frame: 12 months
Measure: Number; unit: percentage probability
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
percentage probability | 81.3

8. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Key Secondary Endpoint: Anatomic Closure of the Primary Target Superficial Truncal Vein at 6 Months.
Description: Anatomic closure of the primary target superficial truncal vein, defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm after VenaSeal™ system and ETA procedures.
  Time to lack of anatomic closure was reported by using the Kaplan-Meier survival probability estimate at 6 months expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of primary target veins with anatomic closure through 6 months.
Time Frame: 6 months
Population: Target Veins based measurement. Number of units analyzed corresponds to the number of primary target veins with data available at the index procedure.
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
Number analyzed (Target Veins) | 131 | 126
percentage probability | 93.9 | 93.5

9. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Key Secondary Endpoint: Anatomic Closure of the Primary Target Superficial Truncal Vein at 6 Months.
Description: Anatomic closure of the primary target superficial truncal vein, defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm after VenaSeal™ system, or the absence of refluxing or residual primary target vein after surgical stripping procedures.
  Time to lack of anatomic closure was reported by using the Kaplan-Meier survival probability estimate at 6 months expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of primary target veins with anatomic closure through 6 months.
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
Number analyzed (Target Veins) | 48 | 43
percentage probability | 97.9 | 92.9

10. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System: Key Secondary Endpoint: Anatomic Closure of the Primary Target Superficial Truncal Vein at 6 Months.
Description: Anatomic closure of the primary target superficial truncal vein, defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm after VenaSeal™ system.
  Time to lack of anatomic closure was reported by using the Kaplan-Meier survival probability estimate at 6 months expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of primary target veins with anatomic closure through 6 months.
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
Number analyzed (Target Veins) | 125
percentage probability | 87.3

11. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Key Secondary Endpoint: Time to Return to Work as Reported by the Patient.
Description: Time to return to work reported by using the cumulative incidence probability estimate of the event happening at 30 days, expressed as a percentage. The data values below represent the cumulative incidence probability as the percentage of participants returning to work through 30 days.
Time Frame: 30 days
Measure: Number; unit: percentage probability
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 94 | 85
percentage probability | 97.9 | 97.6

12. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Key Secondary Endpoint: Time to Return to Work as Reported by the Patient.
Description: as for outcome 11
Time Frame: 30 days
Measure: Number; unit: percentage probability
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 34 | 34
percentage probability | 89.0 | 76.5

13. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System: Key Secondary Endpoint: Time to Return to Work as Reported by the Patient.
Description: as for outcome 11
Time Frame: 30 days
Measure: Number; unit: percentage probability
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 42
percentage probability | 85.7

14. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Anatomic Closure of Primary Target Vein at 30 Days, and 12, 24, 36, 48 and 60 Months.
Description: For subjects treated with the VenaSeal™ system or ETA it is defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm.
  Time to lack of anatomic closure was reported by using the Kaplan-Meier survival probability estimate at 30 days and 12 months, expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of primary target veins with anatomic closure through 30 days and 12 months.
Time Frame: 30 days and 12 months. Data for additional time points 24, 36, 48 and 60 months will be added to additional outcome measure with next posting as data collection is still ongoing.
Population: as for outcome 8
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
Number analyzed (Target Veins) | 131 | 126
percentage probability
  30 days | 95.4 | 95.2
  12 months | 86.6 | 89.3

15. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Anatomic Closure of Primary Target Vein at 30 Days, and 12 Months.
Description: Anatomic closure of the primary target superficial truncal vein, defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm after VenaSeal™ system, or the absence of refluxing or residual primary target vein after surgical stripping procedures.
  Time to lack of anatomic closure was reported by using the Kaplan-Meier survival probability estimate at 30 days and 12 months, expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of primary target veins with anatomic closure through 30 days and 12 months.
Time Frame: 30 days, 12 months
Population: as for outcome 8
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
Number analyzed (Target Veins) | 48 | 43
percentage probability
  30 days | 97.9 | 97.7
  12 months | 95.7 | 92.9

16. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System: Secondary Endpoint: Anatomic Closure of Primary Target Vein at 30 Days, and 12, 24, 36, 48 and 60 Months.
Description: For subjects treated with the VenaSeal™ system it is defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm.
  Time to lack of anatomic closure was reported by using the Kaplan-Meier survival probability estimate at 30 days and 12 months, expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of primary target veins with anatomic closure through 30 days and 12 months.
Time Frame: as for outcome 14
Population: as for outcome 8
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
Number analyzed (Target Veins) | 125
percentage probability
  30 days | 91.9
  12 months | 82.3

17. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Anatomic Closure of Target Vein at 30 Days, and 6, 12, 24, 36, 48 and 60 Months.
Description: For subjects treated with the VenaSeal™ system or ETA this is defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm.
  Time to lack of anatomic closure was reported by using the Kaplan-Meier survival probability estimate at 30 days, 6 months, and 12 months, expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of target veins with anatomic closure through 30 days, 6 months, and 12 months.
Time Frame: 30 days, and 6, 12 months. Data for additional time points 24, 36, 48 and 60 months will be added to additional outcome measure with next posting as data collection is still ongoing.
Population: Target Veins based measurement. Number of units analyzed corresponds to the number of target veins with data available at the index procedure.
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
Number analyzed (Target Veins) | 139 | 132
percentage probability
  30 days | 95.7 | 94.6
  6 months | 93.5 | 93.1
  12 months | 86.6 | 89.0

18. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Anatomic Closure of Target Vein at 30 Days, and 6, 12 Months.
Description: Anatomic closure of target superficial truncal vein defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm after VenaSeal™ system, or the absence of refluxing or residual primary target vein after surgical stripping procedures.
  Time to lack of anatomic closure was reported by using the Kaplan-Meier survival probability estimate at 30 days, 6 months, and 12 months, expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of target veins with anatomic closure through 30 days, 6 months, and 12 months.
Time Frame: 30 days, 6, 12 months
Population: as for outcome 17
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
Number analyzed (Target Veins) | 52 | 45
percentage probability
  30 days | 98.0 | 97.8
  6 months | 98.0 | 93.2
  12 months | 96.0 | 93.2

19. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System: Secondary Endpoint: Anatomic Closure of Target Vein at 30 Days, and 6, 12, 24, 36, 48 and 60 Months.
Description: For subjects treated with the VenaSeal™ system this is defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm.
  Time to lack of anatomic closure was reported by using the Kaplan-Meier survival probability estimate at 30 days, 6 months, and 12 months, expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of target veins with anatomic closure through 30 days, 6 months, and 12 months.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
Number analyzed (Target Veins) | 157
percentage probability
  30 days | 93.6
  6 months | 89.1
  12 months | 85.2

20. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Technical Success of Each Target Vein Immediately Post-index Procedure.
Description: For subjects treated with the VenaSeal™ system or ETA this is defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm.
Time Frame: Post Index procedure, on the day of the procedure immediately following treatment
Population: Target Veins based measurement. Number of units analyzed corresponds to the number of target veins with available data.
Measure: Count of Units; unit: Target Veins
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
Number analyzed (Target Veins) | 138 | 130
Target Veins | 136 | 129

21. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Technical Success of Each Target Vein Immediately Post-index Procedure.
Description: Defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm after VenaSeal™ system, or the absence of refluxing or residual vein after surgical stripping procedures.
Time Frame: Post Index procedure, on the day of the procedure immediately following treatment
Population: Target Veins based measurement. Number of units analyzed corresponds to the number of target veins with available data.
Measure: Count of Units; unit: Target Veins
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
Number analyzed (Target Veins) | 49 | 44
Target Veins | 49 | 44

22. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System: Secondary Endpoint: Technical Success of Each Target Vein Immediately Post-index Procedure.
Description: For subjects treated with the VenaSeal™ system this is defined as DUS showing vein closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm.
Time Frame: Post Index procedure, on the day of the procedure immediately following treatment
Population: Target veins based measurement. Number of analyzed units corresponds to number of target veins with available data.
Measure: Count of Units; unit: Target Veins
Units Other Than Participants: Target Veins
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
Number analyzed (Target Veins) | 153
Target Veins | 147

23. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Reintervention of Any Target Vein (Including Primary Target Vein) Through 12 Months, Assessed at Each Follow-up Visit.
Time Frame: 12 months
Population: Rate based measurement; rate corresponds to count of reinterventions over the total vein-years (sum of patient follow-up time until reintervention, 12 months, or exit if before 12 months, multiplied by number of target veins) among all target veins in the ITT cohort.
Measure: Number; unit: reintervention per vein-years
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 53 | 53
reintervention per vein-years | 0.06 | 0

24. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Time to Reintervention of Any Target Vein (Including Primary Target Vein) Through 12 Months.
Description: As measured by the time between the index procedure and the first reintervention procedure.
  Time to reintervention was reported by using the event free Kaplan-Meier survival probability estimate at 12 months expressed as a percentage. The data values below represent the Kaplan-Meier survival probability as a percentage of target veins without a reintervention through 12 months.
Time Frame: 12 months
Population: Target Veins based measurement. Number of units analyzed corresponds to the number of target veins with available data.
Measure: Number; unit: percentage probability
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
Number analyzed (Target Veins) | 48 | 43
percentage probability | 93.1 | 100

25. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Adverse Events (AEs) Occurring in the Target Limb, Evaluated From Index Procedure Through 12 Months.
Description: Hypersensitivity to VenaSeal™ adhesive, Phlebitis, Granuloma, Endovenous glue induced thrombosis (EGIT) or endovenous heat induced thrombosis (EHIT), Symptomatic deep vein thrombosis (DVT) events.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 136 | 139
Participants
  Hypersensitivity to VenaSeal™ adhesive | 8 | 0
  Phlebitis | 12 | 4
  Granuloma | 1 | 0
  EGIT/EHIT | 1 | 5
  DVT | 0 | 1

26. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Adverse Events (AEs) Occurring in the Target Limb, Evaluated From Index Procedure Through 12 Months.
Description: Hypersensitivity to VenaSeal™ adhesive, Phlebitis, Granuloma, Endovenous glue induced thrombosis (EGIT), Symptomatic deep vein thrombosis (DVT) events.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 53 | 53
Participants
  Hypersensitivity to VenaSeal™ adhesive | 6 | 0
  Phlebitis | 2 | 1
  Granuloma | 0 | 0
  EGIT | 0 | 0
  DVT | 0 | 0

27. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System: Secondary Endpoint: Adverse Events (AEs) Occurring in the Target Limb, Evaluated From Index Procedure Through 12 Months.
Description: as for outcome 26
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
Participants
  Hypersensitivity to VenaSeal™ adhesive | 1
  Phlebitis | 13
  Granuloma | 2
  EGIT | 3
  DVT | 2

28. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Additional Events Evaluated Through 12 Months.
Description: Symptomatic pulmonary embolism (PE), Serious adverse events (SAEs).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 53 | 53
Participants
  Symptomatic pulmonary embolism (PE) | 0 | 0
  Serious adverse events (SAEs) | 1 | 2

29. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Number and Type of Adjunctive Treatments Conducted Through 12 Months Post-index Procedure.
Time Frame: 12 months
Population: Rate based measurement; rate corresponds to the count of adjunctive procedures over the total vein-years (sum of patient follow-up time until adjunct procedure, 12 months, or exit if before 12 months, multiplied by number of target veins) among all target veins in the ITT cohort.
Measure: Number; unit: adjunctive treatment per vein-years
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 136 | 139
Number analyzed (Target Veins) | 144 | 146
adjunctive treatment per vein-years
  Phlebectomy | 0.02 | 0.01
  Sclerotherapy | 0.1 | 0.08

30. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Number and Type of Adjunctive Treatments Conducted Through 12 Months Post-index Procedure.
Time Frame: 12 months
Population: as for outcome 29
Measure: Number; unit: adjunctive treatment per vein-years
Units Other Than Participants: Target Veins
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 53 | 53
Number analyzed (Target Veins) | 59 | 57
adjunctive treatment per vein-years
  Phlebectomy | 0.07 | 0
  Sclerotherapy | 0.07 | 0.02

31. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Number and Type of Adjunctive Treatments Conducted Through 12 Months Post-index Procedure.
Time Frame: 12 months
Population: as for outcome 29
Measure: Number; unit: adjunctive treatment per vein-years
Units Other Than Participants: Target Veins
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
Number analyzed (Target Veins) | 157
adjunctive treatment per vein-years
  Sclerotherapy | 0.12
  Phlebectomy | 0

32. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Healthcare Utilization Related to the Target Limb VRD.
Description: Determined by the number of healthcare visits conducted, and other health-related resources utilized (e.g., home healthcare services) between study visits through 12 months.
Time Frame: 12 months
Population: Rate based measurement; rate corresponds to the count of healthcare utilization over the total person-years (sum of patient follow-up time until Health Care Utilization, 12 months, or exit if before 12 months) among patients in the ITT cohort.
Measure: Number; unit: services utilized per person-years
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 53 | 53
services utilized per person-years
  Inpatient Visits | 0.0210 | 0.0228
  Hospital Outpatient Visits | 0.4409 | 0.1596
  Clinic Visits | 0.0840 | 0.1824
  Outpatient ER Visits | 0.0210 | 0.0228

33. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Procedures, Tests and Treatment of AEs Related to the Treatment Modality or Index Procedure Through 12 Months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 53 | 53
Participants
  Diagnostic Tests Performed: Computed Tomographic Venography | 0 | 0
  Diagnostic Tests Performed: DUS | 4 | 2
  Diagnostic Tests Performed: Intravascular Ultrasound | 0 | 0
  Diagnostic Tests Performed: Magnetic Resonance Venography | 0 | 0
  Diagnostic Tests Performed: Venogram | 0 | 0
  Diagnostic Tests Performed: Other | 1 | 0
  Actions Taken: Medication Change | 9 | 1
  Actions Taken: Intervention Involving Target Limb/Vein | 2 | 2
  Hospitalization | 1 | 1
  Other Actions | 1 | 1

34. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Time to Return to Normal Activities as Reported by the Patients.
Description: Time to return to normal activities reported by using the cumulative incidence probability estimate of the event happening at 30 days, expressed as a percentage. The data values below represent the cumulative incidence probability as the percentage of participants returning to normal activities through 30 days.
Time Frame: 30 days
Measure: Number; unit: percentage probability
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
percentage probability | 98.5 | 96.8

35. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Time to Return to Normal Activities as Reported by the Patients.
Description: as for outcome 34
Time Frame: 30 days
Measure: Number; unit: percentage probability
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
percentage probability | 95.8 | 93.0

36. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Time to Return to Normal Activities as Reported by the Patients.
Description: as for outcome 34
Time Frame: 30 days
Measure: Number; unit: percentage probability
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
percentage probability | 80.9

37. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Intra-procedural and Post-procedural Pain at the Index Procedure, and 7 Days and 30 Days.
Description: Determined by using numeric rating scale (NRS) with a scale of 0-10, with '0' indicating no pain and '10' indicating worst pain imaginable.
Time Frame: Intra-procedure, post-procedure (on the day of the procedure immediately following treatment), 7 days and 30 days
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
score on a scale
  Intra-procedure | 2.0 (2.13) | 2.7 (2.41)
  Post-procedure | 1.1 (1.35) | 1.2 (1.73)
  7 days: number analyzed (Participants) | 127 | 122
  7 days | 1.1 (1.58) | 1.0 (1.40)
  30 days: number analyzed (Participants) | 123 | 115
  30 days | 0.6 (1.05) | 0.7 (1.23)

38. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Intra-procedural and Post-procedural Pain at the Index Procedure, and 7 Days and 30 Days.
Description: as for outcome 37
Time Frame: Intra-procedure, post-procedure (on the day of the procedure immediately following treatment), 7 days and 30 days
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
score on a scale
  Intra-procedure | 1.6 (2.25) | 0.8 (1.95)
  Post-procedure | 1.5 (1.97) | 0.9 (2.00)
  7 days | 2.1 (2.24) | 2.2 (2.10)
  30 days: number analyzed (Participants) | 46 | 43
  30 days | 1.5 (1.92) | 2.3 (2.39)

39. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Intra-procedural and Post-procedural Pain at the Index Procedure, and 7 Days and 30 Days.
Description: as for outcome 37
Time Frame: Intra-procedure, post-procedure (on the day of the procedure immediately following treatment), 7 days and 30 days
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
score on a scale
  Intra-procedure | 3.6 (2.88)
  Post-procedure | 2.3 (2.36)
  7 days: number analyzed (Participants) | 119
  7 days | 2.1 (2.27)
  30 days: number analyzed (Participants) | 119
  30 days | 1.8 (2.32)

40. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Change in Venous Disease Symptoms at 7 and 30 Days, and at 6, 12, 24, 36, 48, and 60 Months Compared to Baseline.
Description: Measured by the revised Venous Clinical Severity Score (rVCSS) and subject self-reporting.
  rVCSS score ranges from 0 to 30, with higher score indicating severe venous disease.
  The outcome measure data reports changes compared to baseline at the different time frames.
Time Frame: 7 and 30 days, and at 6, 12 months. Data for additional time points 24, 36, 48 and 60 months will be added to additional outcome measure with next posting as data collection is still ongoing.
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
score on a scale
  7 days change from baseline: number analyzed (Participants) | 131 | 125
  7 days change from baseline | -2.2 (2.76) | -1.4 (2.51)
  30 days change from baseline: number analyzed (Participants) | 126 | 119
  30 days change from baseline | -3.4 (2.63) | -3.1 (2.70)
  6 months change from baseline: number analyzed (Participants) | 121 | 112
  6 months change from baseline | -4.3 (2.52) | -3.6 (2.84)
  12 months change from baseline: number analyzed (Participants) | 115 | 104
  12 months change from baseline | -3.9 (2.70) | -3.8 (2.93)

41. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Change in Venous Disease Symptoms at 7 and 30 Days, and at 6, 12 Months Compared to Baseline.
Description: as for outcome 40
Time Frame: 7 and 30 days, and at 6 and 12 months
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
score on a scale
  7 days change from baseline | -2.4 (1.90) | -1.6 (2.63)
  30 days change from baseline: number analyzed (Participants) | 46 | 43
  30 days change from baseline | -3.2 (1.78) | -2.2 (2.45)
  6 months change from baseline: number analyzed (Participants) | 41 | 41
  6 months change from baseline | -3.4 (1.79) | -3.0 (2.72)
  12 months change from baseline: number analyzed (Participants) | 43 | 39
  12 months change from baseline | -3.6 (2.16) | -3.6 (2.56)

42. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Change in Venous Disease Symptoms at 7 and 30 Days, and at 6, 12, 24, 36, 48, and 60 Months Compared to Baseline.
Description: as for outcome 40
Time Frame: as for outcome 40
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
score on a scale
  7 days change from baseline: number analyzed (Participants) | 120
  7 days change from baseline | -3.3 (3.96)
  30 days change from baseline: number analyzed (Participants) | 120
  30 days change from baseline | -5.5 (5.01)
  6 months change from baseline: number analyzed (Participants) | 99
  6 months change from baseline | -8.7 (5.27)
  12 months change from baseline: number analyzed (Participants) | 84
  12 months change from baseline | -9.0 (5.44)

43. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Change in AVVQ Score at 30 Days, and 6, 12, 24, 36, 48, and 60 Months Compared to Baseline.
Description: The total score ranges from 0-100 points, with '0' point indicating the best quality of life and '100' points indicating worst quality of life.
  The outcome measure data reports changes compared to baseline at the different time frames.
Time Frame: as for outcome 17
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
score on a scale
  30 days change from baseline: number analyzed (Participants) | 125 | 117
  30 days change from baseline | -5.4 (7.88) | -2.5 (8.19)
  6 months change from baseline: number analyzed (Participants) | 118 | 110
  6 months change from baseline | -7.8 (7.77) | -6.1 (8.88)
  12 months change from baseline: number analyzed (Participants) | 114 | 102
  12 months change from baseline | -8.0 (7.68) | -6.6 (10.37)

44. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Change in AVVQ Score at 30 Days, and 6 and 12 Months Compared to Baseline.
Description: as for outcome 43
Time Frame: 30 days, and 6 and 12 months
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
score on a scale
  30 days change from baseline: number analyzed (Participants) | 45 | 41
  30 days change from baseline | -4.7 (5.94) | -1.0 (8.89)
  6 months change from baseline: number analyzed (Participants) | 40 | 40
  6 months change from baseline | -7.0 (6.26) | -7.7 (7.97)
  12 months change from baseline: number analyzed (Participants) | 41 | 38
  12 months change from baseline | -7.3 (6.13) | -8.8 (6.62)

45. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Change in AVVQ Score at 30 Days, and 6, 12, 24, 36, 48, and 60 Months Compared to Baseline.
Description: as for outcome 43
Time Frame: as for outcome 17
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
score on a scale
  30 days change from baseline: number analyzed (Participants) | 114
  30 days change from baseline | -8.1 (13.67)
  6 months change from baseline: number analyzed (Participants) | 98
  6 months change from baseline | -13.4 (14.40)
  12 months change from baseline: number analyzed (Participants) | 80
  12 months change from baseline | -15.5 (15.21)

46. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Change in EuroQoL Group 5-Dimension Self-Report Questionnaire (EQ-5D-5L) at 30 Days, and 6, 12, 24, 36, 48 and 60 Months Compared to Baseline.
Description: EQ-5D Index scale from <0 to 1.0 (<0 worse than dead, 0 is dead and 1.0 is full health).
  The outcome measure data reports changes compared to baseline at the different time frames.
Time Frame: as for outcome 17
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
score on a scale
  30 days change from baseline: number analyzed (Participants) | 126 | 119
  30 days change from baseline | 0.10 (0.14) | 0.08 (0.15)
  6 months change from baseline: number analyzed (Participants) | 118 | 110
  6 months change from baseline | 0.09 (0.14) | 0.08 (0.18)
  12 months change from baseline: number analyzed (Participants) | 114 | 102
  12 months change from baseline | 0.08 (0.16) | 0.08 (0.15)

47. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Change in EuroQoL Group 5-Dimension Self-Report Questionnaire (EQ-5D-5L) at 30 Days, and 6 and 12 Months Compared to Baseline.
Description: as for outcome 46
Time Frame: 30 days, and 6 and 12 months
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
score on a scale
  30 days change from baseline: number analyzed (Participants) | 46 | 43
  30 days change from baseline | 0.12 (0.19) | 0.15 (0.24)
  6 months change from baseline: number analyzed (Participants) | 40 | 40
  6 months change from baseline | 0.13 (0.19) | 0.13 (0.24)
  12 months change from baseline: number analyzed (Participants) | 42 | 39
  12 months change from baseline | 0.12 (0.22) | 0.14 (0.28)

48. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Change in EuroQoL Group 5-Dimension Self-Report Questionnaire (EQ-5D-5L) at 30 Days, and 6, 12, 24, 36, 48 and 60 Months Compared to Baseline.
Description: as for outcome 46
Time Frame: as for outcome 17
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
score on a scale
  30 days change from baseline: number analyzed (Participants) | 120
  30 days change from baseline | 0.15 (0.24)
  6 months change from baseline: number analyzed (Participants) | 98
  6 months change from baseline | 0.15 (0.25)
  12 months change from basline: number analyzed (Participants) | 84
  12 months change from basline | 0.17 (0.25)

49. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Change in the 36-Item Short Form Health Survey (SF-36) Reported by the Patient at 30 Days, and 6 and 12 Months Compared to Baseline.
Description: The total score ranges from 0 to 100, with higher scores indicating better general health perception.
  The outcome measure data reports changes compared to baseline at the different time frames.
Time Frame: 30 days, and 6 and 12 months
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
score on a scale
  Physical Scale 30 days change from baseline: number analyzed (Participants) | 125 | 117
  Physical Scale 30 days change from baseline | 2.5 (5.86) | 1.8 (5.43)
  Mental Scale 30 days change from baseline: number analyzed (Participants) | 125 | 117
  Mental Scale 30 days change from baseline | 2.1 (9.35) | 0.9 (8.90)
  Physical Scale 6 months change from baseline: number analyzed (Participants) | 117 | 107
  Physical Scale 6 months change from baseline | 2.9 (6.62) | 2.1 (5.46)
  Mental Scale 6 months change from baseline: number analyzed (Participants) | 117 | 107
  Mental Scale 6 months change from baseline | 2.4 (9.77) | 1.3 (8.41)
  Physical Scale 12 months change from baseline: number analyzed (Participants) | 114 | 101
  Physical Scale 12 months change from baseline | 3.1 (6.85) | 1.7 (5.93)
  Mental Scale 12 months change from baseline: number analyzed (Participants) | 114 | 101
  Mental Scale 12 months change from baseline | 2.5 (8.65) | 1.0 (8.28)

50. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Change in the 36-Item Short Form Health Survey (SF-36) Reported by the Patient at 30 Days, and 6 and 12 Months Compared to Baseline.
Description: as for outcome 49
Time Frame: 30 days, and 6 and 12 months
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
score on a scale
  Physical Scale 30 days change from baseline: number analyzed (Participants) | 46 | 43
  Physical Scale 30 days change from baseline | 3.0 (6.50) | 0.5 (6.42)
  Mental Scale 30 days change from baseline: number analyzed (Participants) | 46 | 43
  Mental Scale 30 days change from baseline | 3.4 (9.18) | 2.1 (11.05)
  Physical Scale 6 months change from baseline: number analyzed (Participants) | 40 | 40
  Physical Scale 6 months change from baseline | 3.2 (6.39) | 1.4 (6.15)
  Mental Scale 6 months change from baseline: number analyzed (Participants) | 40 | 40
  Mental Scale 6 months change from baseline | 3.4 (8.21) | 1.6 (8.23)
  Physical Scale 12 months change from baseline: number analyzed (Participants) | 42 | 39
  Physical Scale 12 months change from baseline | 3.7 (7.71) | 2.9 (7.08)
  Mental Scale 12 months change from baseline: number analyzed (Participants) | 42 | 39
  Mental Scale 12 months change from baseline | 1.8 (11.55) | 0.2 (9.71)

51. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Change in the 36-Item Short Form Health Survey (SF-36) Reported by the Patient at 30 Days, and 6 and 12 Months Compared to Baseline.
Description: as for outcome 49
Time Frame: 30 days, and 6 and 12 months
Population: Overall Number of Participants Analyzed is the number of participants that were treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
score on a scale
  Physical Scale 30 days change from baseline: number analyzed (Participants) | 117
  Physical Scale 30 days change from baseline | 2.20 (7.17)
  Mental Scale 30 days change from baseline: number analyzed (Participants) | 117
  Mental Scale 30 days change from baseline | 3.60 (12.13)
  Physical Scale 6 months change from baseline: number analyzed (Participants) | 96
  Physical Scale 6 months change from baseline | 2.86 (7.77)
  Mental Scale 6 months change from baseline: number analyzed (Participants) | 96
  Mental Scale 6 months change from baseline | 5.82 (10.67)
  Physical Scale 12 months change from baseline: number analyzed (Participants) | 83
  Physical Scale 12 months change from baseline | 3.80 (8.23)
  Mental Scale 12 months change from baseline: number analyzed (Participants) | 83
  Mental Scale 12 months change from baseline | 5.81 (11.63)

52. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Change in the Venous Dependent Quality of Life (VenousDQoL) Reported by the Patient at 30 Days, and 6, 12, 24, 36, 48, and 60 Months Compared to Baseline.
Description: Subjects answer their general quality of life with potential responses on an ordinal scale: excellent, very good, good, neither good nor bad, bad, very bad, or extremely bad.
  Subjects also answer what their quality of life would be without varicose veins with potential responses on an ordinal scale: very much better, much better, a little better, the same, or worse.
  The outcome measure data reports the responses at the different time frames including baseline.
Time Frame: as for outcome 17
Population: Overall Number of Participants Analyzed is the number of participants with data at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 122 | 121
Participants
  baseline Quality of Life: Excellent | 16 | 16
  baseline Quality of Life: Very Good | 39 | 32
  baseline Quality of Life: Good | 44 | 49
  baseline Quality of Life: Neither Good Nor Bad | 16 | 17
  baseline Quality of Life: Bad | 7 | 6
  baseline Quality of Life: Very Bad | 0 | 1
  baseline Quality of Life: Extremely Bad | 0 | 0
  baseline Predicted QoL without Varicose Veins: Very Much Better | 32 | 28
  baseline Predicted QoL without Varicose Veins: Much Better | 45 | 42
  baseline Predicted QoL without Varicose Veins: A Little Better | 30 | 37
  baseline Predicted QoL without Varicose Veins: The Same | 15 | 14
  baseline Predicted QoL without Varicose Veins: Worse | 0 | 0
  30 days Quality of Life: Excellent: number analyzed (Participants) | 120 | 115
  30 days Quality of Life: Excellent | 22 | 14
  30 days Quality of Life: Very Good: number analyzed (Participants) | 120 | 115
  30 days Quality of Life: Very Good | 48 | 47
  30 days Quality of Life: Good: number analyzed (Participants) | 120 | 115
  30 days Quality of Life: Good | 40 | 39
  30 days Quality of Life: Neither Good Nor Bad: number analyzed (Participants) | 120 | 115
  30 days Quality of Life: Neither Good Nor Bad | 7 | 11
  30 days Quality of Life: Bad: number analyzed (Participants) | 120 | 115
  30 days Quality of Life: Bad | 3 | 3
  30 days Quality of Life: Very Bad: number analyzed (Participants) | 120 | 115
  30 days Quality of Life: Very Bad | 0 | 1
  30 days Quality of Life: Extremely Bad: number analyzed (Participants) | 120 | 115
  30 days Quality of Life: Extremely Bad | 0 | 0
  30 days Predicted QoL without Varicose Veins: Very Much Better: number analyzed (Participants) | 120 | 115
  30 days Predicted QoL without Varicose Veins: Very Much Better | 28 | 15
  30 days Predicted QoL without Varicose Veins: Much Better: number analyzed (Participants) | 120 | 115
  30 days Predicted QoL without Varicose Veins: Much Better | 30 | 33
  30 days Predicted QoL without Varicose Veins: A Little Better: number analyzed (Participants) | 120 | 115
  30 days Predicted QoL without Varicose Veins: A Little Better | 40 | 31
  30 days Predicted QoL without Varicose Veins: The Same: number analyzed (Participants) | 120 | 115
  30 days Predicted QoL without Varicose Veins: The Same | 22 | 35
  30 days Predicted QoL without Varicose Veins: Worse: number analyzed (Participants) | 120 | 115
  30 days Predicted QoL without Varicose Veins: Worse | 0 | 1
  6 months Quality of Life: Excellent: number analyzed (Participants) | 118 | 110
  6 months Quality of Life: Excellent | 27 | 21
  6 months Quality of Life: Very Good: number analyzed (Participants) | 118 | 110
  6 months Quality of Life: Very Good | 51 | 47
  6 months Quality of Life: Good: number analyzed (Participants) | 118 | 110
  6 months Quality of Life: Good | 35 | 32
  6 Months Quality of Life: Neither Good Nor Bad: number analyzed (Participants) | 118 | 110
  6 Months Quality of Life: Neither Good Nor Bad | 3 | 8
  6 months Quality of Life: Bad: number analyzed (Participants) | 118 | 110
  6 months Quality of Life: Bad | 2 | 1
  6 months Quality of Life: Very Bad: number analyzed (Participants) | 118 | 110
  6 months Quality of Life: Very Bad | 0 | 1
  6 months Quality of Life: Extremely Bad: number analyzed (Participants) | 118 | 110
  6 months Quality of Life: Extremely Bad | 0 | 0
  6 months Predicted QoL without Varicose Veins: Very Much Better: number analyzed (Participants) | 118 | 110
  6 months Predicted QoL without Varicose Veins: Very Much Better | 27 | 17
  6 months Predicted QoL without Varicose Veins: Much Better: number analyzed (Participants) | 118 | 110
  6 months Predicted QoL without Varicose Veins: Much Better | 36 | 27
  6 months Predicted QoL without Varicose Veins: A Little Better: number analyzed (Participants) | 118 | 110
  6 months Predicted QoL without Varicose Veins: A Little Better | 30 | 26
  6 months Predicted QoL without Varicose Veins: The Same: number analyzed (Participants) | 118 | 110
  6 months Predicted QoL without Varicose Veins: The Same | 25 | 39
  6 months Predicted QoL without Varicose Veins: Worse: number analyzed (Participants) | 118 | 110
  6 months Predicted QoL without Varicose Veins: Worse | 0 | 1
  12 months Quality of Life: Excellent: number analyzed (Participants) | 114 | 103
  12 months Quality of Life: Excellent | 24 | 13
  12 months Quality of Life: Very Good: number analyzed (Participants) | 114 | 103
  12 months Quality of Life: Very Good | 49 | 41
  12 months Quality of Life: Good: number analyzed (Participants) | 114 | 103
  12 months Quality of Life: Good | 34 | 36
  12 months Quality of Life: Neither Good Nor Bad: number analyzed (Participants) | 114 | 103
  12 months Quality of Life: Neither Good Nor Bad | 5 | 12
  12 months Quality of Life: Bad: number analyzed (Participants) | 114 | 103
  12 months Quality of Life: Bad | 2 | 1
  12 months Quality of Life: Very Bad: number analyzed (Participants) | 114 | 103
  12 months Quality of Life: Very Bad | 0 | 0
  12 months Quality of Life: Extremely Bad: number analyzed (Participants) | 114 | 103
  12 months Quality of Life: Extremely Bad | 0 | 0
  12 months Predicted QoL without Varicose Veins: Very Much Better: number analyzed (Participants) | 114 | 102
  12 months Predicted QoL without Varicose Veins: Very Much Better | 25 | 14
  12 months Predicted QoL without Varicose Veins: Much Better: number analyzed (Participants) | 114 | 102
  12 months Predicted QoL without Varicose Veins: Much Better | 25 | 27
  12 months Predicted QoL without Varicose Veins: A Little Better: number analyzed (Participants) | 114 | 102
  12 months Predicted QoL without Varicose Veins: A Little Better | 28 | 26
  12 months Predicted QoL without Varicose Veins: The Same: number analyzed (Participants) | 114 | 102
  12 months Predicted QoL without Varicose Veins: The Same | 35 | 34
  12 months Predicted QoL without Varicose Veins: Worse: number analyzed (Participants) | 114 | 102
  12 months Predicted QoL without Varicose Veins: Worse | 1 | 1

53. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Change in the Venous Dependent Quality of Life (VenousDQoL) Reported by the Patient at 30 Days, and 6, 12 Months Compared to Baseline.
Description: as for outcome 52
Time Frame: 30 days, and 6, 12 months
Population: Overall Number of Participants Analyzed is the number of participants with data at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 50 | 47
Participants
  baseline Quality of Life: Excellent | 2 | 2
  baseline Quality of Life: Very Good | 12 | 7
  baseline Quality of Life: Good | 23 | 17
  baseline Quality of Life: Neither Good Nor Bad | 6 | 12
  baseline Quality of Life: Bad | 6 | 4
  baseline Quality of Life: Very Bad | 0 | 1
  baseline Quality of Life: Extremely Bad | 1 | 4
  baseline Predicted QoL without Varicose Veins: Very Much Better | 23 | 18
  baseline Predicted QoL without Varicose Veins: Much Better | 20 | 20
  baseline Predicted QoL without Varicose Veins: A Little Better | 5 | 7
  baseline Predicted QoL without Varicose Veins: The Same | 2 | 2
  baseline Predicted QoL without Varicose Veins: Worse | 0 | 0
  30 days Quality of Life: Excellent: number analyzed (Participants) | 46 | 43
  30 days Quality of Life: Excellent | 5 | 3
  30 days Quality of Life: Very Good: number analyzed (Participants) | 46 | 43
  30 days Quality of Life: Very Good | 17 | 11
  30 days Quality of Life: Good: number analyzed (Participants) | 46 | 43
  30 days Quality of Life: Good | 21 | 20
  30 days Quality of Life: Neither Good Nor Bad: number analyzed (Participants) | 46 | 43
  30 days Quality of Life: Neither Good Nor Bad | 2 | 4
  30 days Quality of Life: Bad: number analyzed (Participants) | 46 | 43
  30 days Quality of Life: Bad | 1 | 3
  30 days Quality of Life: Very Bad: number analyzed (Participants) | 46 | 43
  30 days Quality of Life: Very Bad | 0 | 2
  30 days Quality of Life: Extremely Bad: number analyzed (Participants) | 46 | 43
  30 days Quality of Life: Extremely Bad | 0 | 0
  30 days Predicted QoL without Varicose Veins: Very Much Better: number analyzed (Participants) | 46 | 43
  30 days Predicted QoL without Varicose Veins: Very Much Better | 16 | 15
  30 days Predicted QoL without Varicose Veins: Much Better: number analyzed (Participants) | 46 | 43
  30 days Predicted QoL without Varicose Veins: Much Better | 19 | 24
  30 days Predicted QoL without Varicose Veins: A Little Better: number analyzed (Participants) | 46 | 43
  30 days Predicted QoL without Varicose Veins: A Little Better | 7 | 2
  30 days Predicted QoL without Varicose Veins: The Same: number analyzed (Participants) | 46 | 43
  30 days Predicted QoL without Varicose Veins: The Same | 4 | 2
  30 days Predicted QoL without Varicose Veins: Worse: number analyzed (Participants) | 46 | 43
  30 days Predicted QoL without Varicose Veins: Worse | 0 | 0
  6 months Quality of Life: Excellent: number analyzed (Participants) | 41 | 41
  6 months Quality of Life: Excellent | 7 | 3
  6 months Quality of Life: Very Good: number analyzed (Participants) | 41 | 41
  6 months Quality of Life: Very Good | 17 | 6
  6 months Quality of Life: Good: number analyzed (Participants) | 41 | 41
  6 months Quality of Life: Good | 15 | 23
  6 months Quality of Life: Neither Good Nor Bad: number analyzed (Participants) | 41 | 41
  6 months Quality of Life: Neither Good Nor Bad | 1 | 6
  6 months Quality of Life: Bad: number analyzed (Participants) | 41 | 41
  6 months Quality of Life: Bad | 0 | 1
  6 months Quality of Life: Very Bad: number analyzed (Participants) | 41 | 41
  6 months Quality of Life: Very Bad | 1 | 1
  6 months Quality of Life: Extremely Bad: number analyzed (Participants) | 41 | 41
  6 months Quality of Life: Extremely Bad | 0 | 1
  6 months Predicted QoL without Varicose Veins: Very Much Better: number analyzed (Participants) | 41 | 40
  6 months Predicted QoL without Varicose Veins: Very Much Better | 13 | 15
  6 months Predicted QoL without Varicose Veins: Much Better: number analyzed (Participants) | 41 | 40
  6 months Predicted QoL without Varicose Veins: Much Better | 19 | 17
  6 months Predicted QoL without Varicose Veins: A Little Better: number analyzed (Participants) | 41 | 40
  6 months Predicted QoL without Varicose Veins: A Little Better | 6 | 7
  6 months Predicted QoL without Varicose Veins: The Same: number analyzed (Participants) | 41 | 40
  6 months Predicted QoL without Varicose Veins: The Same | 3 | 1
  6 months Predicted QoL without Varicose Veins: Worse: number analyzed (Participants) | 41 | 40
  6 months Predicted QoL without Varicose Veins: Worse | 0 | 0
  12 months Quality of Life: Excellent: number analyzed (Participants) | 43 | 39
  12 months Quality of Life: Excellent | 8 | 4
  12 months Quality of Life: Very Good: number analyzed (Participants) | 43 | 39
  12 months Quality of Life: Very Good | 16 | 9
  12 months Quality of Life: Good: number analyzed (Participants) | 43 | 39
  12 months Quality of Life: Good | 12 | 15
  12 months Quality of Life: Neither Good Nor Bad: number analyzed (Participants) | 43 | 39
  12 months Quality of Life: Neither Good Nor Bad | 6 | 6
  12 months Quality of Life: Bad: number analyzed (Participants) | 43 | 39
  12 months Quality of Life: Bad | 1 | 5
  12 months Quality of Life: Very Bad: number analyzed (Participants) | 43 | 39
  12 months Quality of Life: Very Bad | 0 | 0
  12 months Quality of Life: Extremely Bad: number analyzed (Participants) | 43 | 39
  12 months Quality of Life: Extremely Bad | 0 | 0
  12 months Predicted QoL without Varicose Veins: Very Much Better: number analyzed (Participants) | 43 | 39
  12 months Predicted QoL without Varicose Veins: Very Much Better | 11 | 12
  12 months Predicted QoL without Varicose Veins: Much Better: number analyzed (Participants) | 43 | 39
  12 months Predicted QoL without Varicose Veins: Much Better | 19 | 17
  12 months Predicted QoL without Varicose Veins: A Little Better: number analyzed (Participants) | 43 | 39
  12 months Predicted QoL without Varicose Veins: A Little Better | 10 | 9
  12 months Predicted QoL without Varicose Veins: The Same: number analyzed (Participants) | 43 | 39
  12 months Predicted QoL without Varicose Veins: The Same | 3 | 1
  12 months Predicted QoL without Varicose Veins: Worse: number analyzed (Participants) | 43 | 39
  12 months Predicted QoL without Varicose Veins: Worse | 0 | 0

54. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Change in the Venous Dependent Quality of Life (VenousDQoL) Reported by the Patient at 30 Days, and 6, 12, 24, 36, 48, and 60 Months Compared to Baseline.
Description: as for outcome 52
Time Frame: as for outcome 17
Population: Overall Number of Participants Analyzed is the number of participants with data at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 123
Participants
  baseline Quality of Life: Excellent | 8
  baseline Quality of Life: Very Good | 21
  baseline Quality of Life: Good | 36
  baseline Quality of Life: Neither Good Nor Bad | 33
  baseline Quality of Life: Bad | 20
  baseline Quality of Life: Very Bad | 4
  baseline Quality of Life: Extremely Bad | 1
  baseline Predicted QoL without Varicose Veins: Very Much Better | 52
  baseline Predicted QoL without Varicose Veins: Much Better | 47
  baseline Predicted QoL without Varicose Veins: A Little Better | 19
  baseline Predicted QoL without Varicose Veins: The Same | 5
  baseline Predicted QoL without Varicose Veins: Worse | 0
  30 days Quality of Life: Excellent: number analyzed (Participants) | 118
  30 days Quality of Life: Excellent | 5
  30 days Quality of Life: Very Good: number analyzed (Participants) | 118
  30 days Quality of Life: Very Good | 36
  30 days Quality of Life: Good: number analyzed (Participants) | 118
  30 days Quality of Life: Good | 42
  30 days Quality of Life: Neither Good Nor Bad: number analyzed (Participants) | 118
  30 days Quality of Life: Neither Good Nor Bad | 24
  30 days Quality of Life: Bad: number analyzed (Participants) | 118
  30 days Quality of Life: Bad | 10
  30 days Quality of Life: Very Bad: number analyzed (Participants) | 118
  30 days Quality of Life: Very Bad | 1
  30 days Quality of Life: Extremely Bad: number analyzed (Participants) | 118
  30 days Quality of Life: Extremely Bad | 0
  30 days Predicted QoL without Varicose Veins: Very Much Better: number analyzed (Participants) | 118
  30 days Predicted QoL without Varicose Veins: Very Much Better | 29
  30 days Predicted QoL without Varicose Veins: Much Better: number analyzed (Participants) | 118
  30 days Predicted QoL without Varicose Veins: Much Better | 58
  30 days Predicted QoL without Varicose Veins: A Little Better: number analyzed (Participants) | 118
  30 days Predicted QoL without Varicose Veins: A Little Better | 20
  30 days Predicted QoL without Varicose Veins: The Same: number analyzed (Participants) | 118
  30 days Predicted QoL without Varicose Veins: The Same | 11
  30 days Predicted QoL without Varicose Veins: Worse: number analyzed (Participants) | 118
  30 days Predicted QoL without Varicose Veins: Worse | 0
  6 Months Quality of Life: Excellent: number analyzed (Participants) | 98
  6 Months Quality of Life: Excellent | 10
  6 Months Quality of Life: Very Good: number analyzed (Participants) | 98
  6 Months Quality of Life: Very Good | 29
  6 Months Quality of Life: Neither Good Nor Bad: number analyzed (Participants) | 98
  6 Months Quality of Life: Neither Good Nor Bad | 16
  6 Months Quality of Life: Good: number analyzed (Participants) | 98
  6 Months Quality of Life: Good | 35
  6 Months Quality of Life: Bad: number analyzed (Participants) | 98
  6 Months Quality of Life: Bad | 6
  6 Months Quality of Life: Very Bad: number analyzed (Participants) | 98
  6 Months Quality of Life: Very Bad | 2
  6 Months Quality of Life: Extremely Bad: number analyzed (Participants) | 98
  6 Months Quality of Life: Extremely Bad | 0
  6 Months Predicted QoL without Varicose Veins: Very Much Better: number analyzed (Participants) | 98
  6 Months Predicted QoL without Varicose Veins: Very Much Better | 27
  6 Months Predicted QoL without Varicose Veins: Much Better: number analyzed (Participants) | 98
  6 Months Predicted QoL without Varicose Veins: Much Better | 35
  6 Months Predicted QoL without Varicose Veins: A Little Better: number analyzed (Participants) | 98
  6 Months Predicted QoL without Varicose Veins: A Little Better | 12
  6 Months Predicted QoL without Varicose Veins: The Same: number analyzed (Participants) | 98
  6 Months Predicted QoL without Varicose Veins: The Same | 24
  6 Months Predicted QoL without Varicose Veins: Worse: number analyzed (Participants) | 98
  6 Months Predicted QoL without Varicose Veins: Worse | 0
  12 Months Quality of Life: Excellent: number analyzed (Participants) | 85
  12 Months Quality of Life: Excellent | 8
  12 Months Quality of Life: Very Good: number analyzed (Participants) | 85
  12 Months Quality of Life: Very Good | 25
  12 Months Quality of Life: Good: number analyzed (Participants) | 85
  12 Months Quality of Life: Good | 30
  12 Months Quality of Life: Neither Good Nor Bad: number analyzed (Participants) | 85
  12 Months Quality of Life: Neither Good Nor Bad | 13
  12 Months Quality of Life: Bad: number analyzed (Participants) | 85
  12 Months Quality of Life: Bad | 7
  12 Months Quality of Life: Very Bad: number analyzed (Participants) | 85
  12 Months Quality of Life: Very Bad | 2
  12 Months Quality of Life: Extremely Bad: number analyzed (Participants) | 85
  12 Months Quality of Life: Extremely Bad | 0
  12 Months Predicted QoL without Varicose Veins: Very Much Better: number analyzed (Participants) | 85
  12 Months Predicted QoL without Varicose Veins: Very Much Better | 19
  12 Months Predicted QoL without Varicose Veins: Much Better: number analyzed (Participants) | 85
  12 Months Predicted QoL without Varicose Veins: Much Better | 22
  12 Months Predicted QoL without Varicose Veins: A Little Better: number analyzed (Participants) | 85
  12 Months Predicted QoL without Varicose Veins: A Little Better | 19
  12 Months Predicted QoL without Varicose Veins: The Same: number analyzed (Participants) | 85
  12 Months Predicted QoL without Varicose Veins: The Same | 24
  12 Months Predicted QoL without Varicose Veins: Worse: number analyzed (Participants) | 85
  12 Months Predicted QoL without Varicose Veins: Worse | 1

55. Secondary Outcome: Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): Secondary Endpoint: Provider Experience Will be Assessed Post-index Procedure, Evaluating Overall Satisfaction With the Procedure.
Description: Measured by a 5 point Likert scale ranging from 0-5, with 5 indicating the best outcome (extremely satisfied with the treatment).
Time Frame: Post-index procedure, on the day of the procedure immediately following treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA
Number analyzed (Participants) | 131 | 126
Participants
  Physician Satisfaction with Procedure: Extremely Satisfied | 77 | 71
  Physician Satisfaction with Procedure: Satisfied | 49 | 52
  Physician Satisfaction with Procedure: Neutral | 4 | 1
  Physician Satisfaction with Procedure: Dissatisfied | 1 | 2
  Physician Satisfaction with Procedure: Extremely Dissatisfied | 0 | 0

56. Secondary Outcome: Randomized Study VenaSeal™ System Versus Surgical Stripping: Secondary Endpoint: Provider Experience Will be Assessed Post-index Procedure, Evaluating Overall Satisfaction With the Procedure.
Description: as for outcome 55
Time Frame: Post-index procedure, on the day of the procedure immediately following treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping
Number analyzed (Participants) | 48 | 43
Participants
  Physician Satisfaction with Procedure: Extremely Satisfied | 10 | 4
  Physician Satisfaction with Procedure: Satisfied | 38 | 27
  Physician Satisfaction with Procedure: Neutral | 0 | 9
  Physician Satisfaction with Procedure: Dissatisfied | 0 | 3
  Physician Satisfaction with Procedure: Extremely Dissatisfied | 0 | 0

57. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Provider Experience Will be Assessed Post-index Procedure, Evaluating Overall Satisfaction With the Procedure.
Description: as for outcome 55
Time Frame: Post-index procedure, on the day of the procedure immediately following treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
Participants
  Physician Satisfaction with Procedure: Extremely Satisfied | 62
  Physician Satisfaction with Procedure: Satisfied | 57
  Physician Satisfaction with Procedure: Neutral | 4
  Physician Satisfaction with Procedure: Dissatisfied | 2
  Physician Satisfaction with Procedure: Extremely Dissatisfied | 0

58. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Peri-procedural Patient Satisfaction as Measured by a Validated Patient-centered Venous Treatment Satisfaction Questionnaire (VenousTSQe) at 30 Days.
Description: as for outcome 1
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 118
score on a scale | 28.2 (6.17)

59. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Patient Satisfaction as Measured by a Validated Patient-centered Venous Treatment Satisfaction Questionnaire (VenousTSQs) at 30 Days.
Description: as for outcome 3
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 118
score on a scale | 30.9 (4.87)

60. Secondary Outcome: Single Arm Venous Leg Ulcer (VLU) Study: Secondary Endpoint: Elimination of Clinically Relevant Superficial Truncal Disease in Target Vein at the Time of Index Procedure as Measured by the Percentage of Target Veins Successfully Treated.
Description: as for outcome 5
Time Frame: Post-index procedure, on the day of the procedure immediately following treatment
Population: Target Veins based measurement. Number of units analyzed corresponds to the number of target veins with available data.
Measure: Mean (Standard Deviation); unit: % of vein length
Units Other Than Participants: Target Veins
Arm/Group | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
Number analyzed (Participants) | 125
Number analyzed (Target Veins) | 153
% of vein length | 90.8 (13.21)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Only adverse events meeting the below criteria will be reported:
  1. All AEs occurring in the target limb, including but not limited to the following specific events:
     * Hypersensitivity
     * Phlebitis
     * Granuloma
     * Endovenous glue induced thrombosis (EGIT) or endovenous heat induced thrombosis (EHIT)
     * Symptomatic DVT.
  2. Symptomatic PEs
  3. Serious adverse events (SAE)
  4. Non-subject (users) adverse events
Arm/Group | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/139 | 0/53 | 0/53 | 10/125
Serious Adverse Events (participants affected / at risk) | 3/136 | 6/139 | 1/53 | 2/53 | 33/125
Other Adverse Events (participants affected / at risk) | 21/136 | 5/139 | 9/53 | 4/53 | 38/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System (N=136) | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA (N=139) | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System (N=53) | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping (N=53) | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System (N=125)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid Mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Cellulitis Staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterobacter Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extradural Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis Infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Streptococcal Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder Mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss Of Personal Independence In Daily Activities (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extremity Necrosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Venous Disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subclavian Vein Occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): VenaSeal™ System (N=136) | Randomized Study VenaSeal™ System Versus Endothermal Ablation (ETA): ETA (N=139) | Randomized Study VenaSeal™ System Versus Surgical Stripping: VenaSeal™ System (N=53) | Randomized Study VenaSeal™ System Versus Surgical Stripping: Surgical Stripping (N=53) | Single Arm Venous Leg Ulcer (VLU) Study: VenaSeal™ System (N=125)
Hypersensitivity (Immune system disorders) | 8 (8) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 25 (28)
Peripheral Venous Disease (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 2 (2)
Phlebitis (Vascular disorders) | 8 (9) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Venous Recanalisation (Vascular disorders) | 5 (5) | 3 (3) | 2 (2) | 0 (0) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT03820947/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03820947/SAP_001.pdf